CLINICAL TRIAL: NCT00033293
Title: A Phase III Randomized Trial of Intravenous Gammaglobulin Therapy for Patients With Neuroblastoma Associated Opsoclonus-Myoclonus-Ataxia Syndrome Treated With Chemotherapy and Prednisone
Brief Title: Cyclophosphamide and Prednisone With or Without Immunoglobulin in Treating Abnormal Muscle Movement in Children With Neuroblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANBL00P3; NCI-2009-00399 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ANBL00P3; CDR0000069271; ANBL00P3 (Other: Children's Oncology Group); ANBL00P3 (Other: CTEP); U10CA013539 (NIH); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-01

CONDITIONS: Localized Resectable Neuroblastoma; Localized Unresectable Neuroblastoma; Regional Neuroblastoma; Stage 4 Neuroblastoma; Stage 4S Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Watchful Waiting; Observation; Cyclophosphamide; Magnetic Resonance Spectroscopy; Prednisone; deltacortene; prednylidene; gamma-Globulins; Immunoglobulins, Intravenous; Immunoglobulins; Antibodies; Panzyga

ARMS (2):
- Arm I (chemotherapy, immunoglobulin therapy) (Experimental): Patients with intermediate-risk or high-risk neuroblastoma receive chemotherapy (including cyclophosphamide) according to the standard of care for the stage of primary neuroblastoma, beginning on day 0. Patients with low-risk neuroblastoma (and not receiving other chemotherapy) receive cyclophosphamide IV over 1 hour on day 0. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. All patients receive oral prednisone twice daily for 3 months and then every other day for 7-15 months.
  Patients receive immune globulin IV on days -2 and -1, at weeks 4, 8, 12, 16, 20, and 24, and then at months 8, 10, and 12 after therapy. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with no response after 6 months go off treatment.
  Interventions: Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Drug: Prednisone; Biological: Therapeutic Immune Globulin
- Arm II (chemotherapy, observation) (Active Comparator): Patients with intermediate-risk or high-risk neuroblastoma receive chemotherapy (including cyclophosphamide) according to the standard of care for the stage of primary neuroblastoma, beginning on day 0. Patients with low-risk neuroblastoma (and not receiving other chemotherapy) receive cyclophosphamide IV over 1 hour on day 0. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. All patients receive oral prednisone twice daily for 3 months and then every other day for 7-15 months.
  Patients do not receive immune globulin. Patients with unresponsive opsoclonus-myoclonus-ataxia syndrome after 2 months or progression after 6 months may cross over to arm I.
  Interventions: Other: Clinical Observation; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Drug: Prednisone

INTERVENTIONS:
Other: Clinical Observation — Undergo observation
  Other Names: observation
  Arms: Arm II (chemotherapy, observation)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Correlative studies
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Drug: Prednisone — Given orally
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Therapeutic Immune Globulin — Given IV
  Other Names: BayGam; Gamimune N; Gamma Globulin; Gammagard S/D; Gammar-P; IgIV; Immune Globulin; Immune Globulin Intravenous; Immune Globulin IV; Iveegam EN; Panglobulin; Panzyga; Polygam S/D; Sandoglobulin; Therapeutic Immunoglobulin; Venoglobulin-I; Venoglobulin-S; WinRho SDF
  Arms: Arm I (chemotherapy, immunoglobulin therapy)

SUMMARY:
This randomized phase III trial is studying cyclophosphamide, prednisone, and immunoglobulin to see how well they work compared to cyclophosphamide and prednisone alone in treating patients with abnormal trunk muscle movements associated with neuroblastoma. Drugs used in chemotherapy, work in different ways to stop tumor cells from dividing so they stop growing or die. Steroid therapy decreases inflammation. Combining chemotherapy and steroid therapy with immunoglobulin may be effective in treating abnormal muscle movement associated with neuroblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether cyclophosphamide and prednisone with or without immune globulin is a reasonable baseline standard therapy for pediatric patients with neuroblastoma-associated opsoclonus-myoclonus-ataxia (OMA) syndrome.

II. Determine whether immunosuppressive therapy with cyclophosphamide and prednisone is an effective backbone therapy for OMA upon which to build additional treatment for these patients

SECONDARY OBJECTIVES:

I. Determine whether these regimens improve OMA syndrome in these patients. II. Determine whether these regimens improve motor coordination in these patients.

III. Determine these regimens improve functional outcome in these patients. IV. Investigate the biology of neuroblastoma associated OMA, with specific regard to magnetic resonance imaging (MRI) findings, anti-neuronal antibodies, cerebrospinal fluid (CSF) findings and tumor biology.

VI. Define better the long-term prognosis for neurologic recovery in the child with neuroblastoma associated with OMA syndrome. VII. Compare the event-free and overall survival of patients treated with these regimens.

OUTLINE:

CHEMOTHERAPY: Patients with intermediate-risk or high-risk neuroblastoma receive chemotherapy (including cyclophosphamide) according to the standard of care for the stage of primary neuroblastoma, beginning on day 0. Patients with low-risk neuroblastoma (and not receiving other chemotherapy) receive cyclophosphamide IV over 1 hour on day 0. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. All patients receive oral prednisone twice daily for 3 months and then every other day for 7-15 months.

IMMUNE GLOBULIN THERAPY: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive immune globulin IV on days -2 and -1, at weeks 4, 8, 12, 16, 20, and 24, and then at months 8, 10, and 12 after therapy. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with no response after 6 months go off treatment.

ARM II: Patients do not receive immune globulin. Patients with unresponsive opsoclonus-myoclonus-ataxia syndrome after 2 months or progression after 6 months may cross over to arm I.

Patients are followed during therapy every month for 6 months, at 1 year, and then annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed neuroblastoma (NBL) or ganglioneuroblastoma with tumor-associated opsoclonus-myoclonus-ataxia syndrome (OMA)

  * Patients with NBL diagnosed within 6 months of OMA diagnosis AND patients with OMA diagnosed within 6 months of NBL diagnosis are eligible
  * Must enroll on study within 4 weeks of diagnosis
  * Presence of opsoclonus, myoclonus, and/or ataxia associated with neuroblastoma considered eligible
* Currently enrolled on COG neuroblastoma protocols: COG-ANBL00B1 or its successor
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR serum creatinine based on age/gender as follows:

  * ≤ 0.4 mg/dL (for patients 1 to 5 months of age)
  * ≤ 0.5 mg/dL (for patients 6 to 11 months of age)
  * ≤ 0.6 mg/dL (for patients 1 year of age)
  * ≤ 0.8 mg/dL (for patients 2 to 5 years of age)
  * ≤ 1.0 mg/dL (for patients 6 to 9 years of age)
  * ≤ 1.2 mg/dL (for patients 10 to 12 years of age)
  * ≤ 1.4 mg/dL (for female patients ≥ 13 years of age)
  * ≤ 1.5 mg/dL (for male patients 13 to 15 years of age)
  * ≤ 1.6 mg/dL (for male patients ≥ 16 years of age)
* No prior IV gamma globulin therapy
* No prior chemotherapy
* Concurrent chemotherapy allowed
* No prior prednisone or corticotropin

  * Patients who have received ≤ 14 days of steroids are eligible
* Concurrent surgery allowed

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2004-03-15 (Actual); Primary Completion 2013-12-10 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro A De Alarcon, Principal Investigator — Children's Oncology Group
Locations (104):
- United States (97):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Harbor-University of California at Los Angeles Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (4):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] de Alarcon PA, Matthay KK, London WB, Naranjo A, Tenney SC, Panzer JA, Hogarty MD, Park JR, Maris JM, Cohn SL. Intravenous immunoglobulin with prednisone and risk-adapted chemotherapy for children with opsoclonus myoclonus ataxia syndrome associated with neuroblastoma (ANBL00P3): a randomised, open-label, phase 3 trial. Lancet Child Adolesc Health. 2018 Jan;2(1):25-34. doi: 10.1016/S2352-4642(17)30130-X. Epub 2017 Nov 3. PMID 29376112
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Chemotherapy, Immunoglobulin Therapy): Patients with intermediate-risk or high-risk neuroblastoma receive chemotherapy (including cyclophosphamide) according to the standard of care for the stage of primary neuroblastoma, beginning day 0. Patients with low-risk neuroblastoma (and not receiving other chemotherapy) receive cyclophosphamide IV over 1 hr on day 0. Treatment repeats every 4 wks for 6 courses in the absence of disease progression or unacceptable toxicity. All patients receive oral prednisone twice daily for 3 mths and then every other day for 7-15 mths.
  Patients receive therapeutic immune globulin IV on days -2 and -1, at wks 4, 8, 12, 16, 20, and 24, and then at mths 8, 10, and 12 after therapy. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with no response after 6 months go off treatment. In case of progression of opsoclonus-myoclonus-ataxia (OMA) during evaluation, patient will be switched to another steroid, corticotropin-releasing hormone (ACTH).
- Arm II (Chemotherapy, Observation): Patients with intermediate-risk or high-risk neuroblastoma receive chemotherapy (including cyclophosphamide) according to the standard of care for the stage of primary neuroblastoma, beginning on day 0. Patients with low-risk neuroblastoma (and not receiving other chemotherapy) receive cyclophosphamide IV over 1 hour on day 0. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. All patients receive oral prednisone twice daily for 3 months and then every other day for 7-15 months.
  Patients do not receive therapeutic immune globulin. Patients with unresponsive opsoclonus-myoclonus-ataxia syndrome after 2 months or progression after 6 months may cross over to arm I.
Period: Overall Study
Arm/Group | Arm I (Chemotherapy, Immunoglobulin Therapy) | Arm II (Chemotherapy, Observation)
Started | 26 | 27
Completed | 16 | 9
Not Completed | 10 | 18
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 5 | 8
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Could not be weaned from steroid therapy | 1 | 1
Not completed — Treatment refused | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Chemotherapy, Immunoglobulin Therapy) | Arm II (Chemotherapy, Observation) | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 27 | 53
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.4 (0.9) | 1.2 (0.5) | 1.3 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 8 | 12 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 19 | 17 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders
Description: A multi-stage design followed by a test of proportions between the treatment arms (chemo vs. chemo + therapeutic immune globulin (IVIG)) will be performed. The first stage of the multi-stage design will also function as an early stopping rule for insufficient activity of chemotherapy in OMA.
Time Frame: Changes from baseline to 2 months, 6 months, and 1 year
Population: Eligible patients
Measure: Number; unit: participants
Arm/Group | Arm I (Chemotherapy, Immunoglobulin Therapy) | Arm II (Chemotherapy, Observation)
Number analyzed (Participants) | 26 | 26
participants | 21 | 11
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, Immunoglobulin Therapy) vs Arm II (Chemotherapy, Observation); The 5 categories of OMA ratings are: stance, gait, arm & hand function, opsoclonus, & mood/behavior. For each category, a patient's response will be based on a comparison of the baseline evaluation to the "best" of 3 time points: 2 months, 6 months & 1 year. If a patient crosses over to the IVIG arm or switches to ACTH at any time, the patient will be considered a non-responder. The proportion of responders from the 2 treatment arms were compared using a chi-squared test; Test type: Other; p = 0.0044, Chi-squared — No adjustments for multiple comparisons; A two-way test with a null hypothesis of no association, using SAS 9.4; Chi-squared test statistic = 8.125

2. Secondary Outcome: Motor Coordination as Assessed by Neurological Examination and Vineland Adaptive Behavior Scale (VABS)
Description: The "best" score at the two time points will be used in this analysis. For a given patient, this "best" score will be used to calculate the change from baseline. The mean change from baseline for each treatment group will be calculated.
Time Frame: Changes from baseline to the better of 6 months or 1 year
Population: All eligible patients who had VABS measures at diagnosis and at least one of 6 months or 1 year.
Measure: Mean (Standard Deviation); unit: Change in VABS score
Groups:
- Arm I (Chemotherapy, Immunoglobulin Therapy): Randomized to chemotherapy, immunoglobulin therapy.
- Arm II (Chemotherapy, Observation): Randomized to chemotherapy, observation
Arm/Group | Arm I (Chemotherapy, Immunoglobulin Therapy) | Arm II (Chemotherapy, Observation)
Number analyzed (Participants) | 17 | 11
Change in VABS score | 84.53 (115.91) | 144.73 (110.69)
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, Immunoglobulin Therapy) vs Arm II (Chemotherapy, Observation); The two samples from the respective treatment arms were compared using a one-sided t-test with a significance level of .05; Test type: Other; p = 0.0919, t-test, 1 sided; Mean Difference (Net) = 60.1979

3. Secondary Outcome: Functional Outcome as Assessed by Age-appropriate Neuropsychological Testing
Description: The Bayley Scales of infant development mental scale "best" score of two time points will be used in the analysis. For a given patient, this score will be used to calculate the change from baseline.
Time Frame: Changes from baseline to the better of 6 months or 1 year
Population: All eligible patients who had Bayley's measures at diagnosis and at least one of 6 months or 1 year.
Measure: Mean (Standard Deviation); unit: Change in Bayley's score
Arm/Group | Arm I (Chemotherapy, Immunoglobulin Therapy) | Arm II (Chemotherapy, Observation)
Number analyzed (Participants) | 4 | 4
Change in Bayley's score | 117.5 (35.35) | 100.75 (25.76)
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, Immunoglobulin Therapy) vs Arm II (Chemotherapy, Observation); Test type: Other — The two samples from the respective treatment arms were compared using a one-sided t-test with a significance level of .05; p = 0.2364, t-test, 1 sided; Mean Difference (Net) = 16.75

4. Secondary Outcome: Biology of Neuroblastoma Associated Opsoclonus-myoclonus-ataxia (OMA) Syndrome Specifically by MRI Findings, Anti-neuronal Antibodies, Cerebrospinal Fluid (CSF) Findings and Tumor Biology
Description: Descriptive analyses on biologic variables will be performed
Time Frame: At diagnosis, 6 months, 1 year, 5 and 10 years after diagnosis
Population: The necessary data will never be collected, therefore results can't be provided.
Arm/Group | Arm I (Chemotherapy, Immunoglobulin Therapy) | Arm II (Chemotherapy, Observation)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Long-term Prognosis for Neurologic Recovery by Neurological Examination
Description: A t-test will be performed on the results of each neurologic test, comparing patients who have had disappearance of anti-neural antibodies to patients whose anti-neural antibodies have not disappeared.
Time Frame: At diagnosis and yearly for 10 years after diagnosis
Population: The necessary data will never be collected, therefore results can't be provided.
Arm/Group | Arm I (Chemotherapy, Immunoglobulin Therapy) | Arm II (Chemotherapy, Observation)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Tumor Outcome in Terms of Event-free Survival (EFS) Rate Defined as a Relapse or Progression of Neuroblastoma, a Second Malignancy, or Death
Description: EFS rate for neuroblastoma event from time of study enrollment.
Time Frame: Up to 3 years
Population: All eligible randomized patients.
Measure: Number (95% Confidence Interval); unit: 3 year EFS
Arm/Group | Arm I (Chemotherapy, Immunoglobulin Therapy) | Arm II (Chemotherapy, Observation)
Number analyzed (Participants) | 26 | 27
3 year EFS | 92.3 [81.8 to 100] | 96.0 [87.8 to 100]

7. Secondary Outcome: Tumor Outcome in Terms of Overall Survival (OS) Rate
Description: OS rate from time of study enrollment.
Time Frame: Up to 3 years
Population: All eligible randomized patients.
Measure: Number (95% Confidence Interval); unit: 3 year OS
Arm/Group | Arm I (Chemotherapy, Immunoglobulin Therapy) | Arm II (Chemotherapy, Observation)
Number analyzed (Participants) | 26 | 27
3 year OS | 100 [100 to 100] | 96.0 [87.8 to 100]

ADVERSE EVENTS:
Description: The SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs), regardless of grade. The other AE field contains all CTCAEs reported on study excluding those that were reported as SAEs, regardless of grade.
Arm/Group | Arm I (Chemotherapy, Immunoglobulin Therapy) | Arm II (Chemotherapy, Observation)
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/27
Other Adverse Events (participants affected / at risk) | 13/26 | 18/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Chemotherapy, Immunoglobulin Therapy) (N=26) | Arm II (Chemotherapy, Observation) (N=27)
53100-Lung infection (Infections and infestations) | 0 (0) | 1 (1)
15000-Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Chemotherapy, Immunoglobulin Therapy) (N=26) | Arm II (Chemotherapy, Observation) (N=27)
13200-Anemia (Blood and lymphatic system disorders) | 1 (3) | 4 (6)
33300-Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (3)
74200-Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
11200-Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
24200-Cushingoid (Endocrine disorders) | 0 (0) | 2 (3)
22100-Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
25700-Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
31200-Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
36700-Gastrointestinal disorders - Other specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
46300-Intra-abdominal hemorrhage(targeted toxicity) (Gastrointestinal disorders) | 0 (0) | 1 (1)
55600-Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
57600-Nausea(targeted toxicity) (Gastrointestinal disorders) | 1 (1) | 2 (5)
87900-Vomiting(targeted toxicity) (Gastrointestinal disorders) | 5 (6) | 5 (10)
33900-Fever (General disorders) | 1 (1) | 1 (1)
48700-Irritability (General disorders) | 0 (0) | 3 (4)
16800-Bladder infection (Infections and infestations) | 2 (2) | 1 (1)
20500-Catheter related infection (Infections and infestations) | 1 (1) | 2 (2)
29500-Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
44800-Infections and infestations - Other specify (Infections and infestations) | 2 (2) | 7 (14)
82300-Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
83100-Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
34900-Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
11600-Alanine aminotransferase increased (Investigations) | 2 (4) | 0 (0)
15000-Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
53700-Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
58300-Neutrophil count decreased (Investigations) | 1 (4) | 3 (8)
65800-Platelet count decreased (Investigations) | 0 (0) | 1 (3)
88200-Weight gain (Investigations) | 0 (0) | 1 (1)
88500-White blood cell decreased (Investigations) | 1 (4) | 2 (3)
13500-Anorexia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
24700-Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
41300-Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
41400-Hyperglycemia(targeted toxicity) (Metabolism and nutrition disorders) | 1 (2) | 4 (6)
41600-Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
42600-Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
42700-Hypocalcemia (Metabolism and nutrition disorders) | 1 (3) | 1 (3)
42900-Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
43100-Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
43300-Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
43500-Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
15300-Ataxia (Nervous system disorders) | 1 (1) | 4 (6)
58700-Nystagmus (Nervous system disorders) | 2 (3) | 9 (14)
69300-Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 1 (1)
11400-Agitation (Psychiatric disorders) | 4 (8) | 11 (25)
13700-Anxiety(targeted toxicity) (Psychiatric disorders) | 0 (0) | 1 (1)
64400-Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
43900-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
41500-Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
69700-Rash maculo-papular(targeted toxicity) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
42100-Hypertension (Vascular disorders) | 0 (0) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval